CLINICAL TRIAL: NCT03091725
Title: Postprandial Nutrient Homeostasis Before and After Weight Loss Induced by Low-calorie Diet or RYGB
Acronym: FGB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Kilo Diabetes & Vascular Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201612107
Record Dates: First submitted 2017-03-13; First posted 2017-03-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Obesity; Roux-en-Y gastric bypass (RYGB); Low calorie diet
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGB group (Experimental): Subjects in this group are scheduled to undergo Roux-en-Y gastric bypass surgery and will be assessed after ~16-18% weight-loss
  Interventions: Procedure: Roux-en-Y gastric bypass surgery
- LCD Group (Active Comparator): Subjects in this group will participate in a low-calorie diet intervention to achieve ~16-18% weight loss.
  Interventions: Behavioral: Low-calorie diet

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass surgery — Roux-en-Y gastric bypass surgery will be performed with post-weight loss testing performed after ~16-18% weight loss is achieved.
  Arms: RYGB group
Behavioral: Low-calorie diet — Subjects will meet with a dietitian and/or behaviorist over 4-6 months to lose ~16-18% of their body weight.
  Arms: LCD Group

SUMMARY:
The purpose of this study is to compare the metabolic responses to low-carbohydrate and standard-carbohydrate meals in African Americans and non-Hispanic White adults with obesity and the effect of weight loss induced by low-calorie diet (LCD) or Roux-en-Y gastric bypass (RYGB) on the metabolic responses to low-carbohydrate and standard meals. Participants will consume: 1) a standard-carbohydrate meal (~49 g glucose) and 2) a low-carbohydrate (~3.4 g glucose) meal on separate study visits performed in a randomized order. We will evaluate the meals' effect before and after ~16-18% weight loss on postprandial i) insulin kinetics, ii) glucose kinetics iii) β-cell function; iv) plasma triglyceride and non-esterified fatty acid concentrations; v) plasma hormone concentrations; vi) plasma cytokine concentrations; vi) plasma metabolomics; and vii) adipose tissue transcriptomics.

ELIGIBILITY:
Inclusion Criteria:

Surgery Group (RYGB):

* Males and Females
* Scheduled for RYGB surgery
* Body Mass Index 35-60 kg/m²
* Without Type 2 Diabetes (T2D)

LCD group:

* Males and Females
* Body Mass Index 35-60 kg/m²
* Without Type 2 Diabetes (T2D)

Exclusion Criteria:

* Regular use of tobacco products
* Previous intestinal resection
* Pregnant or breastfeeding
* Evidence of significant organ system dysfunction or disease other than obesity and T2D
* Use of any medication that might, in the opinion of the investigator, affect metabolic function
* Exercise ≥90 minutes per week
* Use or past use of hormone replacement therapy within the past 6 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Postprandial plasma insulin kinetics | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma insulin kinetics will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial plasma insulin kinetics | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma insulin kinetics will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.

SECONDARY OUTCOMES:
Postprandial glucose kinetics | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma glucose kinetics will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial glucose kinetics | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma glucose kinetics will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
β-cell function | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  β-cell function will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
β-cell function | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  β-cell function will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial triglyceride concentrations | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma triglyceride concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial triglyceride concentrations | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma triglyceride concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial non-esterified fatty acid concentrations | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma non-esterified fatty acid concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial non-esterified fatty acid concentrations | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma non-esterified fatty acid concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial hormone concentrations | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma hormone concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial hormone concentrations | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma hormone concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial cytokine concentrations | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma cytokine concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial cytokine concentrations | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma cytokine concentrations will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal.
Postprandial lipids | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma lipids will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal by using mass spectrometry.
Postprandial lipids | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma lipids will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal by using mass spectrometry.
Postprandial metabolites | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  Plasma metabolites will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal by using mass spectrometry.
Postprandial metabolites | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  Plasma metabolites will be assessed in blood samples collected before and after consuming a standard-carbohydrate or a low-carbohydrate meal by using mass spectrometry.
Transcriptome in adipose tissue | Baseline only (cross-sectional comparison of metabolic responses in African American and non-Hispanic White adults with obesity)
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques in adipose tissue samples collected before and ~3h after consuming a standard-carbohydrate or a low-carbohydrate meal.
Transcriptome in adipose tissue | After 16-18% weight loss induced by LCD or RYGB (~4-6 months)
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques in adipose tissue samples collected before and ~3h after consuming a standard-carbohydrate or a low-carbohydrate meal.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Beth Henk, St Louis, Missouri, United States